CLINICAL TRIAL: NCT00382746
Title: EarlySense Monitoring Device Evaluation on CHF Patients
Status: Withdrawn | Type: Observational
Why Stopped: No need
Sponsor: EarlySense Ltd. (Industry)
Collaborators: Rambam Health Care Campus (Other)
Other Study IDs: ES- CI 02
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-04

CONDITIONS: Congestive Heart Failure
Keywords: Congestive; Heart; Failure; CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: EarlySense monitoring device

SUMMARY:
CHF patients will be monitored using EarlySense ES-16 device and will simultaneously fill diaries and log their weight daily. The data collected and analyzed by the ES-16 device will be correlated with the CHF status data.

ELIGIBILITY:
Inclusion Criteria:

* Age over 45 years old
* CHF class II or III with LVEF<40%
* Hospitalized at least once for CHF deterioration over previous 12 month period
* Able and willing to cooperate with this trial for at least a 3 month period
* Home close to participating center

Exclusion Criteria:

* Recent (within 3 month) admission to ICU or CC-ICU due to severe CHF episode requiring artificial ventilation
* Asthma or COPD

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
CHF | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Rispler, M.D., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel